CLINICAL TRIAL: NCT05924126
Title: Empiric Antibiotic Treatment for Septic Patients in the Intensive Care Unit: Appropriateness and Therapeutic Outcomes
Brief Title: Empiric Antibiotic Treatment for Septic Patients in the Intensive Care Unit
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: MMC-0155-23
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Septic Patients Admitted to the ICU

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- septic patients who recieved appropriate empiric antibiotics
  Interventions: Other: empiric antibiotic therapy
- septic patients who recieved inappropriate empiric antibiotics

INTERVENTIONS:
Other: empiric antibiotic therapy — septic ICU patient given broad spectrum antibiotic therapy
  Groups: septic patients who recieved appropriate empiric antibiotics

SUMMARY:
Sepsis is one of the most common causes of ICU admission. About 5-15% of patients admitted to the hospital with an infection will have sepsis, and about 30-40% of them will have septic shock. About 34% of septic patients and about 53% of patients with septic shock will die within 28 days of admission. Broad-spectrum empiric antibiotic treatment (depending on the source of infection and patient risk factors) is one of the cornerstones of sepsis management. According to the recommendations of the surviving sepsis campaign, empiric antibiotic treatment should be given within one hour of the patient's arrival for patients with sepsis or septic shock. Administration of inappropriate antibiotics in the first 24 hours of admission was found in 34% of septic patients in various studies, and administration of inappropriate antibiotics (or when administered in delay) was found to be associated with increased morbidity and mortality.

In this study, we will assess the proportion of patients who were admitted to the ICU due to sepsis or septic shock and received empiric antibiotic treatment which, in retrospect, according to the growth in the cultures later on, was inappropriate. We will also assess the therapeutic results in these patients - mainly significant morbidity and mortality within 28 days, and compare them to the group of patients who received appropriate antibiotic therapy. We would also like to assess what were the possible reasons for inappropriate empiric antibiotic treatment, in order to draw conclusions to reduce the rate of these cases.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the general ICU due to sepsis or septic shock between 1/1/20 and 31/12/20

Exclusion Criteria: Patients who were admitted due to other non-infectious etiologies

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: septic patients admitted to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of septic patients who recieved inappropriate empiric antibiotic therapy | January 2020-December 2020
  Proportion of septic patients who recieved inappropriate empiric antibiotic therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No